CLINICAL TRIAL: NCT00535262
Title: A Pilot Study Assessing Efficacy, Safety, and Tolerability of EmSam in Bipolar Depression
Brief Title: A Pilot Study Assessing EmSam in Bipolar Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Current lack of medication support.
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #5439
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2014-10-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2013-05

CONDITIONS: Bipolar Depression
Keywords: Bipolar; depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Selegiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EmSam (Experimental): EmSam will be administered in open-label fashion for 8-weeks during phase I of the study during which symptoms of depression will be assessed weekly. Those whose depression responds after 8-weeks will be entered into an 8-month open-label continuation phase during which they will be maintained on EmSam and be assessed on a monthly basis.
  Interventions: Drug: EmSam

INTERVENTIONS:
Drug: EmSam — Selegiline Transdermal System (STS); monoamine oxidase inhibitor patch
  Other Names: Selegiline Transdermal

SUMMARY:
This pilot study will evaluate the efficacy of the monoamine oxidase inhibitor (MAOI)EmSam, a selegiline transdermal system (STS), in bipolar depression.

DETAILED DESCRIPTION:
Most current treatments for bipolar depression have been shown to be of modest effectiveness. There is some literature which suggests that Monoamine Oxidase Inhibitors (MAOIs) have greater efficacy than tricyclic antidepressants, and that they are effective for treatment-resistant depression of all types, both unipolar and bipolar. The MAOI selegiline has demonstrated antidepressant efficacy. EmSam, a selegiline transdermal system, provides central nervous system but not intestinal/liver MAO inhibition without clinically significant increases in sensitivity to dietary tyramine. This transdermal system appears to be associated with fewer side effects and increased safety relative to oral MAOI's. This pilot study will evaluate the efficacy of EmSam in bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 - 65
2. DSM-IV Bipolar Disorder (I, II, NOS), Depressed Phase
3. DSM-IV Bipolar Disorder (I,II, NOS), Mixed state with adequate mood stabilization (ie, resolution of manic or hypomanic symptoms for 8 weeks with a minimum of 4 weeks on a stable dose of mood-stabilizing medication that will be continued through all phases of the study).
4. Prior failure of or inability to tolerate at least one other antidepressant treatment
5. Physically healthy
6. Agrees to participate in the study
7. HAM-D 24 > 10

Exclusion Criteria:

1. Bipolar Disorder (I, II, NOS), Mixed State without adequate mood stabilization
2. Prior significant adverse reaction to EmSam
3. Unstable medical disorder
4. History of epilepsy (febrile seizure o.k.)
5. Current use of any medication that might interact with EnSam.
6. Use within 2 weeks of other antidepressant medication (6 weeks for fluoxetine)
7. Inability to adhere to a tyramine-free diet
8. Recent (past 6 months) suicide attempt
9. Serious suicidal ideation
10. Pregnant
11. Breast feeding
12. Fecund, sexually active females, without adequate contraception
13. Prior failure to respond to 2 or more adequate oral MAOI trials (2/3 PDR maximum dose, minimum 4 weeks)
14. Non-nicotine substance abuse/dependence within the past 6 months (1 year for amphetamines/cocaine)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Deliyannides, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: DES official site — http://www.depression-nyc.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 patients recruited from DES outpatient population with Bipolar Depression, ages 18-65.
Pre-assignment Details: Hypomania/mania requires treatment with mood stabilizer for at least two weeks; must be anti-depressant-free for two weeks (six weeks for fluoxetine.
Groups:
- EmSam: EmSam will be administered in open-label fashion for 8-weeks during phase I of the study during which symptoms of depression will be assessed weekly. Those whose depression responds after 8-weeks will be entered into an 8-month open-label continuation phase during which they will be maintained on EmSam and be assessed on a monthly basis.
  EmSam : Selegiline Transdermal System (STS); monoamine oxidase inhibitor patch
Period: Overall Study
Arm/Group | EmSam
Started | 3 (3 patients were enrolled in the study. Data was collected for only two weeks before funding expired.)
Completed | 0 (Pharmaceutical company withdrew supply of EmSam prematurely before protocol was complete.)
Not Completed | 3
Not completed — No funding | 3

BASELINE CHARACTERISTICS:
Population: Seeking pilot data
Groups:
- Open EmSam: 8-week open-label treatment with EmSam
Arm/Group | Open EmSam
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants] — Patients with Bipolar Depression and one prior anti-depressant treatment with HAM-D (17) score >10 will be entered into treatment.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 3
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Reduction of Depression CGI Score (<= 2)
Description: HAM-D score. Young Mania Scale Life Chart Method Patient Global Impression Symptom Checklist - 90 Quality of Life Enjoyment and Satisfaction Questionnaire
  0 participants analyzed due to early termination of study.
Time Frame: 8 weeks
Groups:
- EmSam: EmSam was administered in open-label fashion during phase I of the study during which symptoms of depression were assessed weekly. The study was terminated early so the data are not reported.
  EmSam : Selegiline Transdermal System (STS); monoamine oxidase inhibitor patch
Arm/Group | EmSam
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | EmSam
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Early termination due to lack of financial support; only 3 participants were entered into the study; no data was analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes